CLINICAL TRIAL: NCT05118646
Title: Comparison of Microcirculation Indexes and Hemodynamic Indexes to Guide Early Fluid Resuscitation in Patients With Septic Shock
Brief Title: Comparison of Microcirculation Indexes and Hemodynamic Indexes to Guide Resuscitation in Patients With Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202006141
Record Dates: First submitted 2021-11-01; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2020-12

CONDITIONS: Sepsis
Keywords: Septic shock; Sublingual Microcirculation
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Hemodynamic Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microcirculation-oriented resuscitation group (Experimental): The microcirculation-oriented resuscitation group will evaluate the organ perfusion level and adjust the hemodynamic therapy according to the sublingual microcirculation parameters (PPV > 68%).
  Interventions: Device: sublingual microcirculation,; Device: hemodynamic monitoring
- Control group (Other): The standard treatment group will adjust the shock management scheme through systemic hemodynamic parameters.
  Interventions: Device: hemodynamic monitoring

INTERVENTIONS:
Device: sublingual microcirculation, — Avoiding pressure artifacts, clear stable microvascular images were taken for a minimum of 20 seconds of the left, middle, and right sections of the tongue.
  Arms: Microcirculation-oriented resuscitation group
Device: hemodynamic monitoring — Arterial blood lactic acid (Lac), central venous oxygen saturation (ScvO2), hematocrit (HCT) and entral venous-to-arterial carbon dioxide partial pressure difference (Pcv-aCO2) will be measured employing a bedside blood gas machine on admission and six hours following admission.

SUMMARY:
Comparison of Microcirculation Indexes and Hemodynamic Indexes to Guide Resuscitation in Patients With Septic Shock

DETAILED DESCRIPTION:
Objectives: Comparison of microcirculation indexes and hemodynamic indexes to guide resuscitation in patients with septic shock.

Intervention:

1. Microcirculation-oriented resuscitation group: When the system hemodynamics meets the standard of EDGT, the microcirculation-oriented resuscitation group will evaluate the organ perfusion level and adjust the hemodynamic therapy according to the sublingual microcirculation parameters (PPV > 68%).
2. Control group: The standard treatment group will adjust the shock management scheme through systemic hemodynamic parameters.

Primary outcome:

(1)change in SOFA score at 72h (2)30-day mortality

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilled the diagnostic criteria of septic shock.

Exclusion Criteria:

* declined to participate
* pregnant
* patients who were younger than 18 years old
* active bleeding
* septic shock is diagnosed for more than 4 hours
* patients are expected to be die within 24hours

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
change in SOFA score | 72h
  △SOFA

SECONDARY OUTCOMES:
30-day mortality | 30d
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: lina Zhang, MD., Principal Investigator — XiangYa Hospital CentralSouth University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China